CLINICAL TRIAL: NCT06139809
Title: The IntubAID Study - Noninvasive Positive Pressure Ventilation During Neonatal Nasal Intubation
Brief Title: Noninvasive Positive Pressure Ventilation During Neonatal Nasal Intubation
Acronym: IntubAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IntubAID
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Infant, Newborn, Diseases; Intubation Complication
Keywords: Intubation; Non-invasive ventilation; Non-invasive positive pressure ventilation; Continuous positive airway pressure; Mechanical ventilation; Physiological stability
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Intubation

STUDY DESIGN:
Intervention Model Description: prospective single-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intubation (Other): Intubation will take place according to our local standard protocol for nasal intubation using non-invasive positive pressure ventilation (NIPPV) delivered through a nasopharyngeal tube. The intubation will be video-recorded to provide a clear view of the procedure and the pulse oximeter displaying the peripheral oxygen saturation (SpO2 [%]) and heart rate (HR [bpm]).
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation — Intubation will take place according to our local standard protocol for nasal intubation using NIPPV delivered through a nasopharyngeal tube. The intubation will be video-recorded to provide a clear view of the procedure and the pulse oximeter displaying the SpO2 and HR.

SUMMARY:
The goal of this study is to perform a quality control assessment of our local intubation protocol in any newborn infant requiring endotracheal intubation in the delivery room or neonatal intensive care unit at the Department of Neonatology of the University Hospital Zurich. The primary aims are:

* Successful nasal intubation at the first attempt without physiological instability.
* Comparison of infants with successful intubation at the first attempt without physiological instability to the infants in the SHINE-Trial in Australia.

Participants will be intubated according to our standard intubation procedure using non-invasive ventilation (NIV) delivered through a nasopharyngeal tube.

ELIGIBILITY:
Inclusion Criteria:

* Any neonate at the Department of Neonatology of the University Hospital Zurich undergoing endotracheal intubation in the delivery room or neonatal intensive care unit.

Exclusion Criteria:

* Requirement for immediate endotracheal intubation as determined by the treating clinician, without time for potential application of NIPPV, e.g. active cardiopulmonary resuscitation.
* Contraindication to NIPPV use (e.g. congenital diaphragmatic hernia, abdominal wall defects).
* Oral intubation planned.
* Denial of parental consent and/or inability of the parents to understand the study procedures due to cognitive or linguistic reasons.
* Withdrawal at the discretion of the intubating clinician if he / she feels the study is interfering with a safe and optimal treatment of the patient.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-31 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
Successful nasal intubation at the first intubation attempt without physiological instability | first intubation attempt
  Number of successful intubations at the first intubation attempt. Physiological instability is defined as the absolute decrease in SpO2 of >20% from baseline and/or bradycardia with a heart rate of <100 bpm for any duration during the first intubation attempt. Baseline is defined as the time immediately before removal of face mask or prong for placement of the nasopharyngeal tube. The intubation starts and ends with the insertion and removal of the laryngoscope blade beyond the infant's lip.

SECONDARY OUTCOMES:
Incidence of desaturation | baseline to begin of first intubation attempt
  Number of desaturations (SpO2 <80 %) between baseline and the begin of the first intubation attempt
Incidence of bradycardia | baseline to begin of first intubation attempt
  Number of bradycardia (HR <100 bpm) between baseline and the begin of the first intubation attempt
Peripheral oxygen saturation | baseline to begin of first intubation attempt
  Mean oxygen saturation over time between baseline and the begin of the first intubation attempt, SpO2 [%]
Heart rate | baseline to begin of first intubation attempt
  Mean heart rate over time between baseline and the begin of the first intubation attempt, HR [bpm]
Incidence of desaturation | first intubation attempt
  Number of desaturations (SpO2 <80 %) during first intubation attempt
Incidence of bradycardia | first intubation attempt
  Number of bradycardia (Hf <100 bpm) during first intubation attempt
Peripheral oxygen saturation | first intubation attempt
  Mean oxygen saturation over time during first intubation attempt, SpO2 [%]
Heart rate | first intubation attempt
  Mean heart rate over time during first intubation attempt, HR [bpm]
Time to desaturation during first intubation attempt | first intubation attempt
  Time [sec] between time zero and desaturation (SpO2 <80%) during the first intubation attempt. Time zero is defined as the time the laryngoscope is inserted past the infant's lips for the first intubation attempt.
Duration of desaturation during first intubation attempt | first intubation attempt
  Time of SpO2 spent below 80% during the first intubation attempt
Time to bradycardia during first intubation attempt | first intubation attempt
  Time [sec] between time zero and bradycardia (HR <100 bpm) during the first intubation attempt.
Duration of bradycardia during first intubation attempt | first intubation attempt
  Time of HR spent below 100 bpm during the first intubation attempt
Duration of intubation attempt(s) | overall intubation procedure
  Time from baseline to successful intubation including all intubation attempts, [sec]
Number of intubation attempts | overall intubation procedure
  Total number of intubation attempts to successful intubation, [n]
Number of disconnections from ventilator circuit | overall intubation procedure
  Total number of disconnections from ventilator circuit between baseline and end of intubation attempt(s), [n]
Incidence of cardiac compressions | Within one hour of first intubation attempt
  Incidence of cardiac compressions within one hour after first intubation attempt, [n]
Incidence of epinephrine administration | Within one hour of first intubation attempt
  Incidence of epinephrine administration within one hour after first intubation attempt, [n]
Incidence of pneumothorax requiring drainage | Within 24 hours of first intubation attempt
  Incidence of pneumothorax requiring drainage within 24 hours after first intubation attempt, [n]
Incidence of death | Within 24 hours of first intubation attempt
  Incidence of death within 24 hours after first intubation attempt, [n]

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bassler, MD, Study Chair — Newborn Research, Depatrment of Neonatology, University Hospital and University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodgson KA, Owen LS, Kamlin COF, Roberts CT, Newman SE, Francis KL, Donath SM, Davis PG, Manley BJ. Nasal High-Flow Therapy during Neonatal Endotracheal Intubation. N Engl J Med. 2022 Apr 28;386(17):1627-1637. doi: 10.1056/NEJMoa2116735. PMID 35476651
- [Background] Kothari R, Hodgson KA, Davis PG, Thio M, Manley BJ, O'Currain E. Time to desaturation in preterm infants undergoing endotracheal intubation. Arch Dis Child Fetal Neonatal Ed. 2021 Nov;106(6):603-607. doi: 10.1136/archdischild-2020-319509. Epub 2021 Apr 30. PMID 33931396
- [Background] Foglia EE, Ades A, Sawyer T, Glass KM, Singh N, Jung P, Quek BH, Johnston LC, Barry J, Zenge J, Moussa A, Kim JH, DeMeo SD, Napolitano N, Nadkarni V, Nishisaki A; NEAR4NEOS Investigators. Neonatal Intubation Practice and Outcomes: An International Registry Study. Pediatrics. 2019 Jan;143(1):e20180902. doi: 10.1542/peds.2018-0902. Epub 2018 Dec 11. PMID 30538147
- [Background] Kamlin CO, O'Connell LA, Morley CJ, Dawson JA, Donath SM, O'Donnell CP, Davis PG. A randomized trial of stylets for intubating newborn infants. Pediatrics. 2013 Jan;131(1):e198-205. doi: 10.1542/peds.2012-0802. Epub 2012 Dec 10. PMID 23230069
- [Background] Lemyre B, Deguise MO, Benson P, Kirpalani H, Ekhaguere OA, Davis PG. Early nasal intermittent positive pressure ventilation (NIPPV) versus early nasal continuous positive airway pressure (NCPAP) for preterm infants. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD005384. doi: 10.1002/14651858.CD005384.pub3. PMID 37466143